CLINICAL TRIAL: NCT04683731
Title: Helping Patients and Providers Make Better Decisions About Colorectal Cancer Screening
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Principal Investigator, Peter Schwartz, Principal Investigator, Indiana University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: 2004109966; CDR-2018C3-14715 (Other Grant/Funding Number: Patient-Centered Outcomes Research Institute)
Record Dates: First submitted 2020-12-20; First posted 2020-12-24 (Actual); Results first posted 2024-12-13 (Actual); Last update posted 2024-12-13 (Actual); Status verified 2024-11

CONDITIONS: Cancer Screening Tests
Keywords: decision aid; cancer screening; risk assessment; risk communication; colorectal neoplasm; decision making
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Decision Support Techniques

STUDY DESIGN:
Intervention Model Description: 2x2, randomized, controlled trial
Who Masked: Participant
Masking Description: Provider-participants will know that their enrolled patient-participant is participating in the study but will not know what arm they were assigned.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group 1 (Active Comparator): Patients view decision aid without personalized message and whose providers do not receive the personalized message.
  Interventions: Behavioral: Decision aid without personalized message; Behavioral: Provider notification without personalized message
- Group 2 (Experimental): Patients view decision aid with personalized message and whose providers do not receive the personalized message.
  Interventions: Behavioral: Decision aid with personalized message; Behavioral: Provider notification without personalized message
- Group 3 (Experimental): Patient view decision aid without the personalized message and whose providers receive the personalized message.
  Interventions: Behavioral: Decision aid without personalized message; Behavioral: Provider notification with personalized message
- Group 4 (Experimental): Patients view decision aid with the personalized message and whose providers receive the personalized message.
  Interventions: Behavioral: Decision aid with personalized message; Behavioral: Provider notification with personalized message

INTERVENTIONS:
Behavioral: Decision aid without personalized message — The decision aid without personalized message consists of a PowerPoint presentation converted to mp4 (video) with text, photos, and an audio track, that is advanced by the viewer and can be viewed online. It begins with a 60 sec video on CRC screening produced by the Centers for Disease Control and Prevention (CDC), followed by slides summarizing the advantages and disadvantages of colonoscopy and stool testing with the fecal immunochemical test (FIT) and DNA+FIT (Cologuard). The presentation is approximately 10 minutes long.
  Arms: Group 1; Group 3
Behavioral: Decision aid with personalized message — The decision aid with personalized message will first present the decision aid without personalized message followed by additional PowerPoint slides converted to mp4 (video) with text, photos, and an audio track briefly explaining the risk tool, the participant's score on the 5 risk factors, total score, ACN risk, and implications for screening and test choice. The presentation is approximately 14 minutes long.
  Arms: Group 2; Group 4
Behavioral: Provider notification without personalized message — Providers will receive a message informing them that their enrolled patient is due for CRC screening. The notification will be sent to them through the electronic health record (EHR) within 24 hours of their visit with the enrolled patient.
  Arms: Group 1; Group 2
Behavioral: Provider notification with personalized message — Providers will receive a message informing them that their enrolled patient is due for CRC screening. The notification will also include the patient's ACN risk (very low, low, moderate, high-average) and implications for screening decisions and test choice. Links to a web landing page containing a more detailed explanation of the risk tool and additional references will be included. The notification will be sent to them through the electronic health record (EHR) within 24 hours of their visit with the enrolled patient.
  Arms: Group 3; Group 4

SUMMARY:
Precision prevention holds great promise for colorectal cancer (CRC) screening but has not been adequately explored. A patient's chance of having an advanced colorectal neoplasm (ACN), i.e. a cancer or precancerous polyp in the colon, significantly affects the comparative effectiveness of approved tests. Giving patients a decision aid with information about their risk for ACN, and giving their providers similar information, could help patients and providers decide if colonoscopy or a non-invasive test (such as the fecal immunochemical test) is more appropriate. This could improve decision making and increase uptake of CRC screening, which are the investigative team's long-term goals.

DETAILED DESCRIPTION:
The research team has developed and pilot tested a decision aid and provider message that discloses the patient's current risk of ACN, based on a prediction rule developed and validated by Dr. Thomas Imperiale, a member of the study team. The Imperiale Prediction Rule uses five variables (gender, age, CRC family history, waist circumference, and smoking history) and identifies a wide range of risk for current ACN among average risk patients. For patients with "high-average" risk (22%), personalized messages in the decision aid and provider notification highlight the advantage of colonoscopy because of the likelihood of finding and removing an ACN. For patients at low risk for ACN (2% or 4%), personalized messages highlight the advantage of stool testing, due to the relatively low chance of failing to detect ACN.

The investigators' long-term goal is to increase uptake of CRC screening by informing and improving patient and provider discussion and decisions. The main objective of this project is to test whether providing patients and their providers with personalized messages about ACN risk results in higher screening uptake and higher decision quality, compared to an approach that does not utilize ACN risk.

ELIGIBILITY:
Inclusion Criteria:

PATIENTS will be eligible if they are:

* age 50 - 75 years
* have not had a colonoscopy performed in the last 10 years, sigmoidoscopy in the last 5 years, fecal occult blood testing (FOBT or FIT) in the last year, or Cologuard in the last 3 years
* have not had a colonoscopy since turning 50 years old
* have a scheduled appointment with a provider who agreed to participate in the study

PROVIDERS will be eligible if they are:

* a physician (MD or DO), nurse practitioner (NP), or physicians assistant (PA) practicing at a partner research site

Exclusion Criteria:

PATIENTS will be excluded if they are:

* undergoing workup for symptoms consistent with CRC, such as unexplained weight loss, change in bowel habit, or rectal bleeding
* have a diagnosis or medical history conferring elevated risk for CRC including a previous adenomatous polyp or CRC, inflammatory bowel disease, high-risk syndromes, or a significant family history of CRC (two or more first degree relatives (FDR) with CRC or one FDR with a CRC diagnosis prior to age 60)
* are unable to speak and read English
* previously participated in any research projects regarding colorectal cancer screening or colonoscopy including, but not limited to the investigators' previous studies
* members of the study team will not be participating in the study; therefore, patients who have a scheduled appointment with any member of the study team will not be eligible.

PROVIDERS will be excluded if they:

* do not have patients between 50 - 75 years old.

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1111 (Actual)
Dates: Start 2021-01-19 (Actual); Primary Completion 2023-05-17 (Actual); Study Completion 2023-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter H. Schwartz, MD, PhD, Principal Investigator — Indiana University
Locations (1):
- Indiana University, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: Yes
Yes, researchers who contact the PI with an IRB-approved protocol may be provided de-identified IPD following our institution's data sharing policies.
Supporting Information: Study Protocol, ICF
Time Frame: Starting in Jan. 2025, indefinitely.
Access Criteria: Contact PI Peter Schwartz (phschwar@iu.edu) and provide IRB-approved protocol for review. Decisions will be made that follow our institution's data sharing policies.

REFERENCES:
- [Derived] Schwartz PH, Perkins SM, Rawl SM, Schmidt KK, Althouse S, Imperiale TF. Effect of Personalized Risk Messages on Uptake of Colorectal Cancer Screening : A Randomized Controlled Trial. Ann Intern Med. 2025 Oct;178(10):1390-1399. doi: 10.7326/ANNALS-24-03144. Epub 2025 Sep 2. PMID 40889370

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited from primary care practices between January 2021 and November 2022.
Groups:
- Group 1: Patients view decision aid without personalized message and whose providers do not receive the personalized message.
  Decision aid without personalized message: The decision aid without personalized message consists of a PowerPoint presentation converted to mp4 (video) with text, photos, and an audio track, that is advanced by the viewer and can be viewed online. It begins with a 60 sec video on CRC screening produced by the Centers for Disease Control and Prevention (CDC), followed by slides summarizing the advantages and disadvantages of colonoscopy and stool testing with the fecal immunochemical test (FIT) and DNA+FIT (Cologuard). The presentation is approximately 10 minutes long.
  Provider notification without personalized message: Providers will receive a message informing them that their enrolled patient is due for CRC screening. The notification will be sent to them through the EHR within 24 hours of their visit with the enrolled patient.
- Group 2: Patients view decision aid with personalized message and whose providers do not receive the personalized message.
  Decision aid with personalized message: The decision aid with personalized message will first present the decision aid without personalized message followed by additional PowerPoint slides converted to mp4 (video) with text, photos, and an audio track briefly explaining the risk tool, the participant's score on the 5 risk factors, total score, advanced colorectal neoplasm (ACN) risk, and implications for screening and test choice. The presentation is approximately 14 minutes long.
  Provider notification without personalized message: Providers will receive a message informing them that their enrolled patient is due for CRC screening. The notification will be sent to them through the EHR within 24 hours of their visit with the enrolled patient.
- Group 3: Patient view decision aid without the personalized message and whose providers receive the personalized message.
  Decision aid without personalized message: The decision aid without personalized message consists of a PowerPoint presentation converted to mp4 (video) with text, photos, and an audio track, that is advanced by the viewer and can be viewed online. It begins with a 60 sec video on CRC screening produced by the Centers for Disease Control and Prevention (CDC), followed by slides summarizing the advantages and disadvantages of colonoscopy and stool testing with the fecal immunochemical test (FIT) and DNA+FIT (Cologuard). The presentation is approximately 10 minutes long.
  Provider notification with personalized message: Providers will receive a message informing them that their enrolled patient is due for CRC screening. The notification will also include the patient's ACN risk (very low, low, moderate, high-average) and implications for screening decisions and test choice. Links to a web landing page containing a more detailed explanation of the risk tool and additional references will be included. The notification will be sent to them through the EHR within 24 hours of their visit with the enrolled patient.
- Group 4: Patients view decision aid with the personalized message and whose providers receive the personalized message.
  Decision aid with personalized message: The decision aid with personalized message will first present the decision aid without personalized message followed by additional PowerPoint slides converted to mp4 (video) with text, photos, and an audio track briefly explaining the risk tool, the participant's score on the 5 risk factors, total score, ACN risk, and implications for screening and test choice. The presentation is approximately 14 minutes long.
  Provider notification with personalized message: Providers will receive a message informing them that their enrolled patient is due for CRC screening. The notification will also include the patient's ACN risk (very low, low, moderate, high-average) and implications for screening decisions and test choice. Links to a web landing page containing a more detailed explanation of the risk tool and additional references will be included. The notification will be sent to them through the EHR within 24 hours of their visit with the enrolled patient.
Period: Overall Study
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4
Started | 294 | 265 | 262 | 290
Completed | 290 | 262 | 247 | 285
Not Completed | 4 | 3 | 15 | 5
Not completed — Withdrawal by Subject | 1 | 0 | 3 | 2
Not completed — Determined patient was not eligible | 3 | 3 | 12 | 3

BASELINE CHARACTERISTICS:
Groups:
- Group 2: Patients view decision aid with personalized message and whose providers do not receive the personalized message.
  Decision aid with personalized message: The decision aid with personalized message will first present the decision aid without personalized message followed by additional PowerPoint slides converted to mp4 (video) with text, photos, and an audio track briefly explaining the risk tool, the participant's score on the 5 risk factors, total score, ACN risk, and implications for screening and test choice. The presentation is approximately 14 minutes long.
  Provider notification without personalized message: Providers will receive a message informing them that their enrolled patient is due for CRC screening. The notification will be sent to them through the EHR within 24 hours of their visit with the enrolled patient.
- Total: Total of all reporting groups
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4 | Total
Number analyzed (Participants) | 290 | 262 | 247 | 285 | 1084
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.2 (5.9) | 56.8 (6.5) | 56.5 (6.2) | 56.4 (6.2) | 56.5 (6.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 173 | 155 | 140 | 179 | 647
  Male | 117 | 107 | 107 | 106 | 437
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Consolidated Race: Black | 76 | 63 | 74 | 77 | 290
  Consolidated Race: Hispanic | 13 | 7 | 8 | 6 | 34
  Consolidated Race: Other | 17 | 15 | 8 | 13 | 53
  Consolidated Race: White | 171 | 165 | 148 | 180 | 664
  Consolidated Race: Unknown or Not Reported | 13 | 12 | 9 | 9 | 43
Region of Enrollment [Number; unit: participants]
  United States | 290 | 262 | 247 | 285 | 1084
Education - highest level [Count of Participants; unit: Participants]
  Less than high school | 9 | 16 | 10 | 10 | 45
  High school graduate/GED | 45 | 54 | 55 | 55 | 209
  Some college or technical school/trade school | 79 | 67 | 59 | 68 | 273
  Associates degree | 28 | 32 | 24 | 26 | 110
  Bachelors degree | 69 | 42 | 53 | 68 | 232
  Professional or graduate degree | 38 | 33 | 29 | 45 | 145
  Prefer not to answer | 9 | 6 | 6 | 5 | 26
  Unknown or Not Reported | 13 | 12 | 11 | 8 | 44
Relationship [Count of Participants; unit: Participants]
  Divorced | 69 | 46 | 54 | 62 | 231
  Married or living with a partner | 140 | 141 | 128 | 144 | 553
  Never married | 43 | 43 | 40 | 43 | 169
  Separated | 14 | 7 | 9 | 10 | 40
  Widowed | 12 | 13 | 7 | 17 | 49
  Unknown or Not Reported | 12 | 12 | 9 | 9 | 42
Employed? [Count of Participants; unit: Participants]
  Yes | 183 | 165 | 147 | 172 | 667
  No | 95 | 85 | 89 | 105 | 374
  Unknown or Not Reported | 12 | 12 | 11 | 8 | 43
Health Insurance? [Count of Participants; unit: Participants]
  Yes | 268 | 241 | 228 | 264 | 1001
  No | 10 | 9 | 9 | 13 | 41
  Unknown or Not Reported | 12 | 12 | 10 | 8 | 42
Insurance Lapse over 12 Months? [Count of Participants; unit: Participants]
  Yes | 27 | 12 | 24 | 24 | 87
  No | 238 | 227 | 200 | 239 | 904
  Unknown or Not Reported | 25 | 23 | 23 | 22 | 93
Self-reported Health Status at Baseline [Count of Participants; unit: Participants]
  Excellent | 10 | 10 | 10 | 16 | 46
  Very Good | 59 | 52 | 50 | 70 | 231
  Good | 121 | 117 | 104 | 114 | 456
  Fair | 74 | 62 | 58 | 64 | 258
  Poor | 12 | 9 | 15 | 13 | 49
  Missing or Not Reported | 14 | 12 | 10 | 8 | 44
Subjective Income Level [Count of Participants; unit: Participants]
  Are comfortable | 124 | 134 | 114 | 126 | 498
  Have just enough to make ends meet | 109 | 93 | 86 | 108 | 396
  Do NOT have enough to make ends meet | 41 | 23 | 36 | 42 | 142
  Missing or Not Reported | 16 | 12 | 11 | 9 | 48
Subjective Numeracy [Mean (Standard Deviation); unit: units on a scale] — Subjective numeracy was assesses using the short, 3-item version of the Subjective Numeracy Scale, a validated instrument that involves Likert-type questions regarding the participant's preference for or dislike of numeric information and their perception of their ability to understand it. Each item has a six-point response option from 1-6. A mean across the three items was calculated and the mean could range from 1 to 6. A higher score means the participant has a greater preference for numeric information and/or greater perception of their ability to understand numeric information.
  units on a scale | 4.2 (1.3) | 4.3 (1.2) | 4.2 (1.3) | 4.3 (1.2) | 4.3 (1.3)
Health Literacy [Mean (Standard Deviation); unit: units on a scale] — The Health Literacy Scale, a 3-item scale, was used. Scores were summed to obtain a total score. Scores can range from 0-12 and a higher score indicates lower health literacy.
  units on a scale | 2.1 (2.4) | 1.9 (2.2) | 2.1 (2.2) | 1.9 (2.2) | 2.0 (2.3)
Perceived Comparative Risk for Colorectal Cancer [Count of Participants; unit: Participants] — Perceived Comparative Colorectal Cancer (CRC) Risk was assessed with a single item which asked "compared to other women/men your same age, would you say your chance of getting colon cancer in the next 10 years is higher, about the same, lower, or don't know.
  Participants
    Lower than other women/men your age | 68 | 54 | 53 | 73 | 248
    About the same as other women/men your age | 111 | 101 | 101 | 110 | 423
    Higher than other women/men your age | 13 | 7 | 15 | 9 | 44
    Don't know | 88 | 92 | 72 | 86 | 338
    Unknown or Not Reported | 10 | 8 | 6 | 7 | 31

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Completed Colorectal Cancer Screening
Description: Patients' completion of colonoscopy, fecal immunochemical testing (FIT), or other CRC screening within 6 months, based on documentation in the participants' electronic health record.
Time Frame: 6 months after patient enrollment
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4
Number analyzed (Participants) | 290 | 262 | 247 | 285
Participants | 110 | 95 | 113 | 113

2. Primary Outcome: Number of Participants Who Made a High Quality Decision Using the Multi-dimensional Measure of Informed Consent (MMIC) Which Incorporates Knowledge, Intent, and Behavior.
Description: Decision quality will be assessed using the multi-dimensional measure of informed consent (MMIC), where a high-quality decision is one where the individual has adequate knowledge regarding the available options and undergoes the screening test that he or she has chosen or that fits his or her values ("values concordance"). Patient knowledge of colorectal cancer and screening will be assessed by a 12-item test made up of 6 multiple choice questions and 6 true-false questions. Adequate knowledge = 9 correct. Concordance will be measured between the patient's test choice at the post-provider survey and the screening test underwent, if any, within 6 months after patient enrollment.
Time Frame: 6 months after participant enrollment
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4
Number analyzed (Participants) | 290 | 262 | 247 | 285
Participants | 90 | 92 | 91 | 103

3. Secondary Outcome: Number of Participants Who Completed Colorectal Cancer Screening by Type of Screening Test Completed
Description: Colorectal cancer (CRC) screening uptake and type of screening test completed within 6 months of enrolled was assessed, as documented in the electronic health record (EHR).
Time Frame: 6 months after participant enrollment
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4
Number analyzed (Participants) | 290 | 262 | 247 | 285
Participants
  Completed a colonoscopy | 59 | 39 | 52 | 51
  Completed a stool test (FIT or Cologuard) | 51 | 56 | 61 | 62
  Did not complete a CRC screening test | 180 | 167 | 134 | 172

4. Secondary Outcome: Average Intention to Get a Colorectal Cancer (CRC) Screening Test of Participants: Change Between Baseline, Post-intervention, and Post-provider Visit
Description: Patients' intention to be screened for CRC with any CRC screening test will be measured with 1 item: "Do you plan to get any type of colon cancer screening test within the next 6 months?". The response options were: 5=Definitely; 4=Probably; 3=May or may not; 2=Probably not; and 1=Definitely not. Higher positive change means CRC screening intention increased. Increased intention to be screened is a better outcome.
Time Frame: 1 day (immediately before viewing intervention [baseline/T1] and after viewing intervention [post-intervention/T1]); and approximately 4-30 days after viewing intervention and 4-14 days after provider visit (post-provider visit/T2)
Population: Only participants who completed the item at each time point under comparison were used in the analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4
Number analyzed (Participants) | 290 | 262 | 247 | 285
score on a scale
  Change from baseline (T0) to post-intervention (T1): number analyzed (Participants) | 267 | 246 | 225 | 268
  Change from baseline (T0) to post-intervention (T1) | 0.59 (0.79) | 0.68 (0.86) | 0.55 (0.84) | 0.63 (0.83)
  Change from post-intervention (T1) to post-provider visit (T2): number analyzed (Participants) | 220 | 198 | 187 | 230
  Change from post-intervention (T1) to post-provider visit (T2) | 0.23 (0.93) | 0.24 (0.74) | 0.24 (0.82) | 0.20 (0.79)
  Change from baseline (T0) to post-provider visit (T2): number analyzed (Participants) | 224 | 204 | 197 | 235
  Change from baseline (T0) to post-provider visit (T2) | 0.85 (1.18) | 0.94 (1.01) | 0.80 (1.15) | 0.82 (1.05)

5. Secondary Outcome: Number of Participants Intended Colorectal Cancer (CRC) Screening Behavior
Description: For those patients who answer the screening intent item with "definitely not," "probably not," or "may or may not", test choice will be categorized as "no screening". Those who answer Screening Intent with "Probably" or "Definitely" have Test Choice categorized based on their answer to a single item: "If you have a colon test, which one would you choose?" Response options are: Stool test (FIT or Cologuard), Colonoscopy, Another test, or Don't know.
Time Frame: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4
Number analyzed (Participants) | 290 | 262 | 247 | 285
Participants
  Intended screening behavior at baseline (T0): Intends to be screened with colonoscopy | 70 | 58 | 56 | 79
  Intended screening behavior at baseline (T0): Intends to be screened with a stool test (FIT or Cologuard) | 62 | 53 | 55 | 70
  Intended screening behavior at baseline (T0): Intends to be screened with another test | 2 | 3 | 2 | 2
  Intended screening behavior at baseline (T0): Intends to be screened and don't know which test | 37 | 37 | 35 | 32
  Intended screening behavior at baseline (T0): Does not intend to be screened | 111 | 105 | 95 | 99
  Intended screening behavior at baseline (T0): Unknown or not reported | 8 | 6 | 4 | 3
  Intended screening behavior at post-intervention (T1): Intends to be screened with colonoscopy | 106 | 82 | 93 | 86
  Intended screening behavior at post-intervention (T1): Intends to be screened with a stool test (FIT or Cologuard) | 85 | 106 | 74 | 133
  Intended screening behavior at post-intervention (T1): Intends to be screened with another test | 0 | 0 | 1 | 0
  Intended screening behavior at post-intervention (T1): Intends to be screened and don't know which test | 25 | 18 | 19 | 19
  Intended screening behavior at post-intervention (T1): Does not intend to be screened | 52 | 40 | 39 | 31
  Intended screening behavior at post-intervention (T1): Unknown or not reported | 22 | 16 | 21 | 16
  Intended screening behavior at post-provider (T2): Intends to be screened with colonoscopy | 104 | 90 | 83 | 89
  Intended screening behavior at post-provider (T2): Intends to be screened with a stool test (FIT or Cologuard) | 92 | 84 | 89 | 117
  Intended screening behavior at post-provider (T2): Intends to be screened with another test | 1 | 1 | 0 | 1
  Intended screening behavior at post-provider (T2): Intends to be screened and don't know which test | 6 | 5 | 2 | 3
  Intended screening behavior at post-provider (T2): Does not intend to be screened | 26 | 25 | 25 | 27
  Intended screening behavior at post-provider (T2): Unknown or not reported | 61 | 57 | 48 | 48

6. Secondary Outcome: Average Correct Responses of Participants to Knowledge Questions About Colorectal Cancer (CRC) and CRC Screening: Change Between Baseline, Post-intervention, and Post-provider Visit.
Description: Knowledge was assessed with six multiple choice and six true/false questions regarding general information (including risk factors, screening test options, and test frequency) of CRC and CRC screening. Knowledge scores were derived by summing correct responses to the 12 individual knowledge questions (range, 0-12), and change was calculated from baseline (T0) to post-intervention (T1), post-intervention (T1) to post-provider visit (T2), and from baseline (T0) to post-provider (T2) by using the knowledge score at the later time point minus the knowledge score of the former time point. The range for change could be -12 to 12 with higher values meaning an increase in knowledge which is a better outcome.
Time Frame: as for outcome 4
Population: Only participants who completed the item at each time point under comparison were used in the analysis.
Measure: Mean (Standard Deviation); unit: units on a scale-number correct
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4
Number analyzed (Participants) | 290 | 262 | 247 | 285
units on a scale-number correct
  Change in correct responses from baseline (T0) to post-intervention (T1): number analyzed (Participants) | 267 | 244 | 222 | 263
  Change in correct responses from baseline (T0) to post-intervention (T1) | 3.65 (2.68) | 3.70 (2.74) | 3.75 (2.82) | 3.76 (2.90)
  Change in correct responses from post-intervention (T1) to post-provider visit (T2): number analyzed (Participants) | 219 | 197 | 183 | 225
  Change in correct responses from post-intervention (T1) to post-provider visit (T2) | -0.60 (1.40) | -0.58 (1.31) | -0.60 (1.60) | -0.43 (1.45)
  Change in correct responses from baseline (T0) to post-provider visit (T2): number analyzed (Participants) | 224 | 204 | 194 | 231
  Change in correct responses from baseline (T0) to post-provider visit (T2) | 3.03 (2.71) | 3.10 (2.79) | 3.02 (3.02) | 3.31 (2.83)

7. Secondary Outcome: Average Perceived Personal Colorectal Cancer Risk of Participants: Change Between Baseline, Post-intervention, and Post-provider Visit
Description: Multiple choice questions assessing the patients' perception of how likely they are to get colon cancer in the next 5 years, in the next 10 years, and sometime during their lifetime. Each has response options: 4=very likely, 3=somewhat likely, 2=somewhat unlikely, and 1=very unlikely. The mean of the 3 questions was calculated (each combined score has a range of 1 to 4) at each time point. We calculated the change from baseline (T0) to post-intervention (T1), post-intervention (T1) to post-provider visit (T2), and from baseline (T0) to post-provider (T2) by using the mean of the later time point minus the mean of the former time point.
  The range for change could be from -3 to 3 with higher values meaning an increase in perceived risk.
Time Frame: as for outcome 4
Population: Only participants who completed the item at each time point under comparison were used in the analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4
Number analyzed (Participants) | 267 | 244 | 223 | 264
score on a scale
  Change from baseline (T0) to post-intervention (T1) | 0.21 (0.74) | 0.15 (0.78) | 0.14 (0.81) | 0.08 (0.77)
  Change from post-intervention (T1) to post-provider visit (T2): number analyzed (Participants) | 219 | 197 | 184 | 225
  Change from post-intervention (T1) to post-provider visit (T2) | -0.10 (0.86) | 0.12 (0.82) | 0.10 (0.87) | 0.05 (0.83)
  Change from baseline (T0) to post-provider visit (T2): number analyzed (Participants) | 224 | 203 | 196 | 231
  Change from baseline (T0) to post-provider visit (T2) | 0.14 (0.79) | 0.28 (0.87) | 0.21 (0.98) | 0.14 (0.84)

8. Secondary Outcome: Average Decision Conflict of Participants: Change Between Baseline, Post-intervention, and Post-provider Visit
Description: Patients' decision conflict is assessed using the low literacy version of the Decision Conflict Scale, a ten-item instrument that assesses patients' subjective feeling regarding the decision process over five areas. Each item has three response categories (yes, no, unsure). Scores are summed; divided by 10; and multiplied by 25. Scores range from 0 [no decisional conflict] to 100 [extremely high decisional conflict]. Negative change means decision conflict decreased. A decrease in decision conflict is a better outcome.
Time Frame: as for outcome 4
Population: Only participants who completed the item at each time point under comparison were used in the analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4
Number analyzed (Participants) | 267 | 244 | 222 | 263
score on a scale
  Change from baseline (T0) to post-intervention (T1) | -36.6 (28.9) | -42.4 (27.6) | -37.1 (27.7) | -40.3 (28.4)
  Change from post-intervention (T1) to post-provider visit (T2): number analyzed (Participants) | 219 | 197 | 183 | 225
  Change from post-intervention (T1) to post-provider visit (T2) | -1.60 (12.1) | -0.76 (9.53) | -2.32 (11.6) | -0.27 (11.6)
  Change from baseline (T0) to post-provider visit (T2): number analyzed (Participants) | 224 | 204 | 196 | 230
  Change from baseline (T0) to post-provider visit (T2) | -39.0 (29.2) | -41.6 (28.8) | -37.9 (29.2) | -39.3 (29.2)

9. Secondary Outcome: Number of Participants Who Perceive Being Involved in Shared-Decision Making as Assessed by the Shared Decision Making Process Survey-4
Description: Patients answered four items assessing the extent to which they were involved in the decision-making process. Each item had response options: 1= A lot; 2=Some; 3=A little; 4=Not at all. Each item was analyzed separately and responses "A lot", "Some" and "A little" were considered "enough" and received 1 point. The response "Not at all" was considered "not enough" and received 0 points.
Time Frame: approximately 4-30 days after viewing intervention and 4-14 days after provider visit [post-provider visit/T2]
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4
Number analyzed (Participants) | 290 | 262 | 247 | 285
Participants
  How much did you and your provider talk about the reasons you might want to have a colonoscopy?: Enough | 203 | 178 | 164 | 201
  How much did you and your provider talk about the reasons you might want to have a colonoscopy?: Not enough | 26 | 28 | 35 | 35
  How much did you and your provider talk about the reasons you might want to have a colonoscopy?: Unknown or not reported | 61 | 56 | 48 | 49
  How much did you and your provider talk about the reasons you might not want to have a colonoscopy?: Enough | 106 | 89 | 91 | 119
  How much did you and your provider talk about the reasons you might not want to have a colonoscopy?: Not enough | 123 | 117 | 108 | 117
  How much did you and your provider talk about the reasons you might not want to have a colonoscopy?: Unknown or not reported | 61 | 56 | 48 | 49
  How much did you and your provider talk about the reasons you might want to do a stool test?: Enough | 160 | 146 | 146 | 173
  How much did you and your provider talk about the reasons you might want to do a stool test?: Not enough | 69 | 60 | 52 | 63
  How much did you and your provider talk about the reasons you might want to do a stool test?: Unknown or not reported | 61 | 56 | 49 | 49
  How much did you and your provider talk about the reasons you might not want to do a stool test?: Enough | 108 | 92 | 93 | 111
  How much did you and your provider talk about the reasons you might not want to do a stool test?: Not enough | 121 | 114 | 106 | 124
  How much did you and your provider talk about the reasons you might not want to do a stool test?: Unknown or not reported | 61 | 56 | 48 | 50

10. Secondary Outcome: Number of Participants Who Perceive Being Involved in Shared-Decision Making as Assessed by the Decision Quality Instrument
Description: A single-item measure taken from the Colon Cancer Testing Decision Quality Worksheet v.2.0 assessing if the patients' primary care provider asked them which type of colon cancer screening test they wanted.
Time Frame: approximately 4-30 days after viewing intervention and 4-14 days after provider visit [post-provider visit/T2]
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4
Number analyzed (Participants) | 290 | 262 | 247 | 285
Participants
  Yes | 152 | 134 | 130 | 159
  No | 76 | 72 | 69 | 77
  Unknown or not reported | 62 | 56 | 48 | 49

11. Secondary Outcome: Participant's Average Perception of Shared-Decision Making as Assessed by CollaboRATE
Description: A 3-item measure assessing how much effort was made by their provider to: explain colon cancer screening, ask for screening preferences, and incorporate those preferences into the decision. Response options ranged from 0="No effort was made" to 9="Every effort was made". The three items were summed and a mean was calculated. Scores can range from 0-9. A higher score indicates more perceived shared decision making. Higher perceived shared decision making is a better outcome.
Time Frame: approximately 4-30 days after viewing intervention and 4-14 days after provider visit [post-provider visit/T2]
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4
Number analyzed (Participants) | 290 | 262 | 247 | 285
score on a scale | 6.4 (3.1) | 6.3 (3.2) | 6.3 (3.2) | 6.5 (3.0)

12. Secondary Outcome: Number of Participants With Orders for a Colorectal Cancer Screening (CRC) Test
Description: A FIT, colonoscopy, or other CRC screening test ordered within 6 months of each participants' enrollment based on documentation in the electronic health record (EHR).
Time Frame: 6 months after patient enrollment
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4
Number analyzed (Participants) | 290 | 262 | 247 | 285
Participants
  NO order for CRC screening test | 89 | 84 | 79 | 84
  YES order for CRC screening test | 201 | 178 | 168 | 201

13. Secondary Outcome: Number of Providers Who Open Their Provider Notification
Description: Opening the provider notification sent for each patient was assessed by reviewing the electronic health record (EHR).
Time Frame: 6 months after patient enrollment
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4
Number analyzed (Participants) | 290 | 262 | 247 | 285
Participants
  Provider notification was opened | 181 | 161 | 153 | 175
  Provider notification was not opened | 34 | 33 | 29 | 28
  Provider notification was not sent | 7 | 4 | 7 | 2
  Unable to determine if provider notification was opened | 68 | 64 | 58 | 80

ADVERSE EVENTS:
Time Frame: 28 months
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4
All-Cause Mortality (participants affected / at risk) | 0/290 | 0/262 | 0/247 | 0/285
Serious Adverse Events (participants affected / at risk) | 0/290 | 0/262 | 0/247 | 0/285
Other Adverse Events (participants affected / at risk) | 0/290 | 0/262 | 0/247 | 0/285

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-05-01): https://cdn.clinicaltrials.gov/large-docs/31/NCT04683731/Prot_SAP_000.pdf